CLINICAL TRIAL: NCT07316868
Title: Neuroprotective Effect of Mild Hypothermia as Compared With Normothermia During Cardiopulmonary Bypass of Coronary Artery Bypass Grafting - A Single-center Randomized Controlled Trial
Brief Title: Neuroprotective Effect of Mild Hypothermia Versus Normothermia During Cardiopulmonary Bypass of Coronary Artery Surgery
Acronym: HYPNOCABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Timo Laitio, Professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VARHA/4272/13.02.02/2025
Record Dates: First submitted 2025-11-24; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Brain Injury
Keywords: hypothermia; normothermia; cardiopulmonary bypass; coronary artery bypass grafting; diffusion tensor imaging; neuroprotection; biomarkers
MeSH Terms: conditions — Coronary Artery Disease; Brain Injuries; Hypothermia

STUDY DESIGN:
Intervention Model Description: This is a single-blinded randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Intervention group: normothermic cardiopulmonary bypass with nasopharyngeal temperature of 36.5 ± 0.2°C
  Interventions: Procedure: Normothermic cardiopulmonary bypass
- Control group (Active Comparator): Control group: mild hypothermic cardiopulmonary bypass with nasopharyngeal temperature of 33 ± 0.2°C
  Interventions: Procedure: Hypothermic cardiopulmonary bypass

INTERVENTIONS:
Procedure: Normothermic cardiopulmonary bypass — normothermic cardiopulmonary bypass with nasopharyngeal temperature of 36.5 ± 0.2°C
  Other Names: 36.5 ± 0.2°C
  Arms: Intervention group
Procedure: Hypothermic cardiopulmonary bypass — mild hypothermic cardiopulmonary bypass with nasopharyngeal temperature of 33 ± 0.2°C
  Other Names: 33 ± 0.2°C
  Arms: Control group

SUMMARY:
In high-income countries, coronary artery bypass grafting (CABG) remains a common procedure, with approximately 36.7 operations per 100,000 inhabitants annually, corresponding to about 136,000 procedures in the European Union. This highlights the substantial healthcare burden and the need to optimize surgical outcomes. Cardiopulmonary bypass (CPB) is a fundamental component of cardiac surgery, ensuring extracorporeal perfusion of vital organs.

Hypothermic CPB has historically been widely used for organ protection due to its presumed neuroprotective mechanisms. However, evidence demonstrating its superiority over normothermic CPB remains inconclusive. In its 2024 guidelines, the European Association for Cardio-Thoracic Surgery recommends considering normothermia (≥35 °C) to reduce postoperative neurocognitive dysfunction (Class II, Level A). This recommendation is primarily based on two meta-analyses, but the underlying studies show methodological heterogeneity, outdated practices, and limited applicability to contemporary cardiac surgery. Importantly, the guidelines acknowledge the need for large randomized controlled trials to define optimal target temperature management (TTM) during CPB.

Previous diffusion-weighted MRI studies have demonstrated silent ischemic brain lesions in approximately 30% of CABG patients, with postoperative neurocognitive decline occurring in a similar proportion. However, no significant differences have been shown between normothermic and hypothermic CPB. Diffusion tensor imaging (DTI) extends conventional diffusion imaging by enabling detailed assessment of white matter microstructure and tractography. Fractional anisotropy (FA), a key DTI metric, has demonstrated prognostic value in various neurological conditions but has not yet been applied in CABG patients.

Blood-based biomarkers, including glial fibrillary acidic protein, neurofilament light chain, neuron-specific enolase, and total tau, offer complementary insights into brain injury but have not been studied in combination with DTI in this population.

This study will compare mild hypothermic (33-34 °C) and normothermic (36.5 °C) CPB to evaluate their neuroprotective effects using advanced MRI techniques and blood-based biomarkers. The primary aim is to determine whether mild hypothermia provides superior neuroprotection following CABG. Secondary objectives include assessing white matter injury evolution, global ischemic burden, associations with biomarkers and neurocognitive decline, and developing integrated prognostic models to improve outcomes in CABG patients.

DETAILED DESCRIPTION:
In high-income countries, 36.7 coronary artery bypass grafting (CABG) procedures are performed per 100,000 population each year, translating to approximately 136,000 procedures in the European Union, and thereby underscoring the significant healthcare burden and importance of optimizing surgical outcomes. During cardiac surgery, cardiopulmonary bypass (CPB), a cornerstone of cardiac surgery, ensures extracorporeal perfusion to critical organs.

Historically, hypothermic CPB has been employed in the majority of cardiac operations and remains one of the most common methods for organ protection in routine cardiac surgery. The biological rationale for hypothermia is grounded in its multiple mechanisms of neuroprotection. Despite these findings, the superiority of hypothermic CPB over normothermic CPB in terms of neuroprotection remains uncertain.

In its 2024 guidelines, the European Association for Cardio-Thoracic Surgery recommends considering normothermia (defined as temperatures ≥ 35°C) to reduce the risk of postoperative neurocognitive dysfunction (Class II, Level A recommendation). Hypothermia, in this context, is defined as a core temperature below 35°C. The recommendation is based on two recent meta-analyses: Abbasciano et al. 2022 and Linassi et al. 2022. However, the 2024 recommendation is underpinned by evidence that remains limited in quality and relevance. The key studies included in these meta-analyses exhibit methodological inconsistencies and rely on outdated definitions and clinical practices, thereby limiting the generalizability and applicability of the findings to current cardiac surgical and anesthetic practice. Notably, the recommendation itself acknowledges the need for large randomized controlled trials to determine the optimal target temperature management (TTM) during cardiopulmonary bypass (CPB).

Previous studies using diffusion-weighted imaging (DWI) in magnetic resonance imaging (MRI) have revealed silent ischemic brain lesions, predominantly deep white matter lesions, in approximately 30% of patients following CABG. Furthermore, postoperative neurocognitive decline occurs in an average of 30.2% of CABG patients. However, earlier DWI and neurocognitive studies have not demonstrated statistically significant differences between normothermic and hypothermic CPB.

Diffusion tensor imaging (DTI) extends the capabilities of DWI and offers several advantages. Unlike DWI, which measures diffusion magnitude, DTI provides detailed quantitative insights into white matter architecture and allows for visualization and quantification of white matter tracts through tractography. Fractional anisotropy (FA), a key DTI parameter, quantifies the magnitude and directionality of water diffusion within white matter tracts. FA has shown independent prognostic value for neurological outcomes in patients with traumatic brain injury, subarachnoid hemorrhage, or cardiac arrest. Despite its potential, DTI has not yet been applied to CABG patients. This technique could significantly enhance our understanding of white matter microintegrity evolution and overall injury burden following CABG, insights necessary for optimizing TTM during CPB.

In addition to brain imaging with DTI, blood-based biomarkers such as glial fibrillary acidic protein (GFAP), neurofilament light chain (NfL), neuron-specific enolase (NSE), and total tau (T-tau) provide complementary tools for monitoring brain injury progression and improving prognostication of long-term neurological outcomes. Each biomarker are expressed in different cellular origins and exhibit distinct characteristics and temporal dynamics, potentially offering unique insights into the extent of brain injury post-CABG. However, their ability to independently or synergistically measure white and gray matter injury in combination with DTI parameters remains unexplored in CABG patients.

To optimize TTM during CPB, this study will investigate the neuroprotective effects of hypothermic (33-34 °C) and normothermic (36.5 °C) CPB by evaluating their impact on white matter injury, cerebral perfusion, and whole-brain neural networks using advanced MRI techniques.

The primary aim of this study is to evaluate whether mild hypothermic CPB offers superior neuroprotection compared to normothermic CPB. This will be assessed using brain DTI and blood-based biomarkers following CABG. Secondary objectives include evaluating the evolution of white matter architecture, the extent of global ischemic injury to white matter microintegrity, and the association between these factors, postoperative blood-based biomarker levels, and neurocognitive decline. In addition, an objective is to develop innovative and highly precise prognostic models by integrating advanced brain imaging technologies with comprehensive biomarker analysis. Ultimately, the overarching goal is to identify factors that can improve the treatment outcomes for patients undergoing CABG.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained
2. Age of >18 years
3. Undergoing elective or subacute coronary artery bypass grafting

Exclusion Criteria:

1. An emergency case
2. A history of stroke
3. A history of intracranial bleeding
4. A history of transient ischemic attack (TIA)
5. A history of neurodegenerative diseases such as Alzheimer's, multiple sclerosis
6. The subject is known to have a clinically significant laboratory abnormality, medical condition (such as decompensated liver disease or severe chronic obstructive pulmonary disease), or social circumstance that, in the investigator's opinion, makes it inappropriate for the subject to participate in this clinical trial.
7. Presence of implants or foreign bodies which are not known to be MRI safe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Global fractional anisotropy of brain white matter of diffusion tensor imaging (DTI) | Postoperative Day 6 +/- 1 day
  Fractional anisotropy measures white matter microintegrity. It is assessed with brain magnetic resonance diffusion tenson imaging (DTI)

SECONDARY OUTCOMES:
Change in hippocampal volume in milliliters (ml) from preoperative day 4 (+/- 3 days) to postoperative day 6 (+/-1 day) between the control and the intervention group | Change of hippocampal volume between preoperative day 4 +/- 3 days and postoperative day 6 +/- 1day
  The volume of hippocampus will be measured with voxel-based morphometry of magnetic resonance imaging at preoperative day 4 +/- 3 days and at postoperative day 6 +/- 1day.
Number of participants with treatment related adverse events as assessed by CTCAE v 4.0 | From enrollment to the end of follow-up at 1 year
Change in hippocampal ischemic injury from preoperative day 4 +/- 3 days to postoperative day 6 +/- 1 day between the control group and the intervention group. | The change of hippocampal ischemic injury from the preoperative day 4 +/-3 days to postoperative day 6 +/- 1 day
  The ischemic injury in the hippocampus will be measured with magnetic resonance diffusion tensor imaging
Change in ischemic injury of basal ganglia from preoperative day 4 +/- 3 days to postoperative day 6+/- 1 day between the control group and the intervention group | The change of ischemic injury in basal ganglia from the ppreoperative day 4 +/- 3 days to postoperative day 6 +/- 1 day
  The ischemic injury in basal ganglia will be measured with the magnetic resonance diffusion tensor imaging
Change of global white matter injury as assessed with diffusion tensor imaging between the control group and the intervention group from preoperative day 4 +/- 3 days to postoperative day 6 +/- 1 day and to 3 months +/- 7 days | Change of global ischemic white matter injury from preoperative day 4 +/- 3 to postoperative day 6 +/-1 day and to 3 months +/- 7 days
  The global (i.e. the whole brain) ischemic white matter injury will be measured with fractional anisotropy and with radial, axial and mean diffusivity of the magnetic resonance diffusion tensor imaging. These parameters are always measured simultaneously and cannot be separated.
Change of global gray matter injury between the control group and the intervention group from preoperative day 4 +/- 3 days to postoperative day 6 +/- 1 day and to 3 months +/- 7 days | Change of global gray matter injury from preoperative day 4 +/- 3 days to postoperative day 6 +/- 1 day and to 3 months +/- 7 days after operation
  The global (i.e. the whole brain) gray matter injury will be measured with mean diffusivity of diffusion tensor imaging
Difference of blood-based neuron specific enolase (NSE) between the control group and the intervention group | NSE is analysed immediately prior to anesthesia induction and at postoperative 24, 48 and at 72 hours
  NSE is analyzed from a blood sample
Difference of blood-based neurofilament light chain (NfL) between the control group and the intervention group | NfL is analyzed immediately prior to anesthesia induction and at postoperative 24, 48 and at 72 hours
  NfL is analyzed from a blood sample
Difference of blood-based glial fibrillary acidic protein (GFAP) between the control group and the intervention group | GFAP is analyzed immediately prior to anesthesia induction and at postoperative 24, 48 and at 72 hours
  GFAP is analyzed from a blood sample
Difference of blood-based total tau between the control group and the intervention group | total tau is analyzed immediately prior to anesthesia induction and at postoperative 24, 48 and at 72 hours
  total tau is analyzed from a blood sample
Difference of neurocognitive outcomes between the control group and the intervention group as assessed with the Cambridge Neuropsychological Test Automated Battery (CANTAB) | CANTAB will be assessed at preoperative day 2 +/- 1 day and postoperatively at 3 and at 12 months
Difference of intraoperative Near-Infrared Spectroscopy NIRS values between the control and the intervention group during . | NIRS will be measured intraoperatively
Difference in the need for vasoactive medication between the control group and the intervention group. | 96 hours after start of anesthesia induction
  Vasoactive medication includes norepinephrine, epinephrine, vasopressin, levosimendan and nitroglycerin
The need for antipyretic medication between the contorl group and the interventin group | 96 hours after start of anesthesia induction
Blood lactate levels between the control group and the intervention group | Lactate will be measured intraoperatively at 1-hour intervals and at intervals of 2 to 6 hours from the start to the end of postoperative intensive care
Difference of a quantity of blood products and hemostatic agents between the control and the intervention group | 96 hours after start of anesthesia induction
Difference of the length of intensive care unit stay between the control group and the intervention group | 96 hours after start of anesthesia induction

CONTACTS AND LOCATIONS:
Overall Officials: Timo Laitio, MD, PhD, Principal Investigator — Turku University Hospital, Wellbeing Services County of Southwest Finland
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
Primary endpoint
Supporting Information: CSR
Time Frame: from January 1, 2027 to December 31, 2029
Access Criteria: The data of this study will be available to investigators whose proposed use of the data has been approved by an independent review committee. Individual participant data that underlie the results reported in this Article will be shared (text, tables, figures, and appendices), after de-identification, along with the study protocol. These data will be available 6 months after the Article's publication and will be available for 12 months from publication. Data can be used for individual participant data meta-analysis. Requests and proposals should be directed to timo.laitio@elisanet.fi. To gain access, data requestors will need to sign a data access agreement.